CLINICAL TRIAL: NCT05633680
Title: Detection of Folate Receptor-positive Circulating Tumor Cells as a Biomarker for Diagnosis
Brief Title: Circulating Tumor Cells Screen for Breast Cancer
Acronym: CTCSFBC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Handan First Hospital (Other)
Responsible Party: Principal Investigator, kunwu-yan, Research Project Leader, Handan First Hospital
Other Study IDs: handan1; 20200187 (Other Grant/Funding Number: 2020 Hebei Provincial Health Commission Youth Project Fund Project)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasm; Neoplastic Cells, Circulating
Keywords: Breast cancer; Circulating tumor cells
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast cancer group: Breast cancer is finally determined through breast puncture biopsy or excisional tissue biopsy and sent for pathological diagnosis
  Interventions: Diagnostic Test: Peripheral blood sampling for circulating tumor cells
- Non-breast cancer group: By breast puncture biopsy or excisional tissue biopsy and sent to pathology for final determination of benign tumor. and healthy women
  Interventions: Diagnostic Test: Peripheral blood sampling for circulating tumor cells

INTERVENTIONS:
Diagnostic Test: Peripheral blood sampling for circulating tumor cells — Patients had 3-4 ml of venous blood drawn on day 1 after admission, ethylene diamine tetra acetic acid (EDTA) was used for anticoagulation, samples were stored at 4 ℃, and CTCs analysis was performed within 24 hours after collection. .FU/3 ml was used as the unit for CTC quantification.

SUMMARY:
A prospective study was used to collect patients considering breast cancer admitted to our general surgery department from 2019-6 to 2023-8, to identify the case group (breast cancer) and the control group (non-breast cancer), to compare the differences in CTC in peripheral blood between the two groups, and to draw conclusions after statistical analysis.

DETAILED DESCRIPTION:
This project is a prospective study by collecting clinical data from breast cancer and non-breast cancer patients admitted to our general surgery department from 2020 to 2023, and drawing peripheral blood for CTC testing. The clinical data of 200 patients were initially collected and grouped, with the study group positioned as breast cancer patients (patients with pathologically determined breast cancer) and the control group as non-breast cancer patients (patients with benign breast tumors and healthy women), to investigate the expression of CTC in breast cancer and correlation with the degree of metastasis, as well as to further understand the relationship between CTC in peripheral blood and breast cancer clinicopathology. The circulating tumor cell enrichment was compared between the two groups, and the data were derived for statistical analysis to draw conclusions, as well as to identify shortcomings and make improvements to the existing problems.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of breast cancer Must be able to cooperate with the examination

Exclusion Criteria:

patients were currently undergoing or had prior cancer treatment; patients had other conditions which investigators thought not suitable for the study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with a clinical diagnosis of breast cancer, patients with benign breast disease (BBD), and healthy females were recruited for this study, Patients with benign breast disease and healthy women as negative controls.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Enrichment of circulating tumor cells | 1 week
  The main test was the enrichment of circulating tumor cells in the peripheral blood of the two groups of patients.FU/3 ml was used as the unit for CTC quantification.

CONTACTS AND LOCATIONS:
Overall Officials: kunwu yan, Master, Principal Investigator — Handan First Hospital
Locations (1):
- Kunwu Yan, Handan, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Chen C, Ke J, Zhou XE, Yi W, Brunzelle JS, Li J, Yong EL, Xu HE, Melcher K. Structural basis for molecular recognition of folic acid by folate receptors. Nature. 2013 Aug 22;500(7463):486-9. doi: 10.1038/nature12327. Epub 2013 Jul 14. PMID 23851396
- [Background] Haber DA, Velculescu VE. Blood-based analyses of cancer: circulating tumor cells and circulating tumor DNA. Cancer Discov. 2014 Jun;4(6):650-61. doi: 10.1158/2159-8290.CD-13-1014. Epub 2014 May 6. PMID 24801577
- [Background] Sparano J, O'Neill A, Alpaugh K, Wolff AC, Northfelt DW, Dang CT, Sledge GW, Miller KD. Association of Circulating Tumor Cells With Late Recurrence of Estrogen Receptor-Positive Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1700-1706. doi: 10.1001/jamaoncol.2018.2574. PMID 30054636
- [Background] Goodman CR, Seagle BL, Friedl TWP, Rack B, Lato K, Fink V, Cristofanilli M, Donnelly ED, Janni W, Shahabi S, Strauss JB. Association of Circulating Tumor Cell Status With Benefit of Radiotherapy and Survival in Early-Stage Breast Cancer. JAMA Oncol. 2018 Aug 1;4(8):e180163. doi: 10.1001/jamaoncol.2018.0163. Epub 2018 Aug 9. PMID 29800954
- [Background] Banko P, Lee SY, Nagygyorgy V, Zrinyi M, Chae CH, Cho DH, Telekes A. Technologies for circulating tumor cell separation from whole blood. J Hematol Oncol. 2019 May 14;12(1):48. doi: 10.1186/s13045-019-0735-4. PMID 31088479